CLINICAL TRIAL: NCT03291431
Title: Intermittent Theta Burst TMS for the Treatment of Alcohol Use Disorders in Veterans
Brief Title: Intermittent Theta Burst for the Treatment of Alcohol Use Disorders in Veterans
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties due to Covid-19 pandemic
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Timothy Durazzo, PhD, Associate Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 41896
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Results first posted 2023-06-22 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Alcohol Use Disorder; Depressive Disorder; Cigarette Smoking
Keywords: alcohol use disorder; intermittent theta burst; Veterans; depressive disorder; cigarette smoking
MeSH Terms: conditions — Alcoholism; Depressive Disorder; Cigarette Smoking

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Active iTBS (Active Comparator): Participants will be randomized to active or sham iTBS.
  Interventions: Device: Intermittent theta burst transcranial magnetic stimulation
- Sham iTBS (Sham Comparator): Participants will be randomized to active or sham iTBS.
  Interventions: Device: Intermittent theta burst transcranial magnetic stimulation

INTERVENTIONS:
Device: Intermittent theta burst transcranial magnetic stimulation — 20 iTBS sessions (active or sham) administered over the course of 2 weeks

SUMMARY:
The purpose of this study is to evaluate the efficacy of intermittent theta burst repetitive transcranial magnetic stimulation (iTBS) as a treatment for Veterans with an alcohol use disorder (AUD) to decrease the exceedingly high rate of relapse associated with this condition. iTBS has demonstrated equivalent efficacy and safety to repetitive transcranial magnetic stimulation employing 10Hz stimulation protocols in treatment of depressive disorders. The advantage of iTBS is that it can be delivered in approximately 5 minutes where conventional 10Hz repetitive transcranial magnetic stimulation (rTMS) protocols are typically 20-25 minutes. It is hypothesized that Veterans with AUD who receive active iTBS applied to the left dorsolateral prefrontal cortex (DLPFC), compared to controls (i.e., Veterans with AUD who receive sham iTBS), will show significant decreases alcohol craving, depressive symptomatology and cigarette consumptions, as well as improved neurocognition, a longer period of abstinence, and a lower overall rate of relapse over 6 months following standard psychosocial treatment for AUD at VA substance treatment clinics. In exploratory analyses, it is also predicted that magnetic resonance measures of left DLPFC glutamate concentration, volume of anterior frontal cortical brain regions, and performance on fMRI tasks interrogating the function of the salience/reward circuits will serve as biomarkers of iTBS treatment response. The goal of this proposal is to implement treatment that effectively promotes sustained abstinence in Veterans with AUD, given long-term abstinence is related to optimal neurobiological, neuropsychological and psychosocial recovery and functioning.

ELIGIBILITY:
Inclusion Criteria:

* 21-65 years of age
* Meet Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) criteria for alcohol use disorder, and alcohol is self-identified as primary substance of misuse.
* Actively in treatment at VA Palo Alto HCS Addiction Treatment Service
* Able to read, verbalize understanding, and voluntarily sign the Informed Consent Form prior to participation in study procedures.

Exclusion Criteria:

* History of Schizophrenia Spectrum Disorders, Bipolar Disorders, a
* Current substance use disorder that exceeds the severity of the AUD (based on DSM-5 diagnostic criteria)
* Current use of an FDA approved medication (i.e., disulfiram, acamprosate, and naltrexone) for treatment of AUD,
* Active current suicidal intent or plan (patients with a previous clinical flag for risk for suicide will be required to have an established safety plan involving their primary psychiatrist and the treatment team before entering the clinical trial),
* Any form of previous TMS or electroconvulsive treatment.
* Thyroid disease,
* Unstable congestive heart failure, angina, other severe cardiac illness as defined by treatment regimen changes in the prior 3 months
* Cerebrovascular accident
* Cancer if < 1 year since end of treatment
* Unstable diabetes
* COPD requiring oxygen supplementation
* Alzheimer's disease
* Parkinson's disease
* Any Biomedical implants with ferromagnetic content
* Neurostimulation devices, cardiac pacemakers or any magnetic resonance contraindications
* Traumatic brain injury with self-reported or observed loss of consciousness > 30 minutes
* Any primary or traumatically induced seizure disorder
* Lack of fluency in English, Wechsler Adult Reading Test below the 7th percentile (i.e., moderate or greater impairment in estimated general intelligence),
* Females who are pregnant or actively attempting pregnancy (conservative exclusion for magnetic resonance research),
* Current use of any medication or substance that is documented to lower seizure threshold or has been identified as a contraindication for TMS treatment.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-07-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Timothy C Durazzo, PhD, Principal Investigator — Stanford University
Locations (2):
- United States (2):
  - Palo Alto VA Health Care System, Palo Alto, California
  - Stanford University, Stanford, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Durazzo TC, McNerney MW, Hansen AM, Gu M, Sacchet MD, Padula CB. BDNF rs6265 Met carriers with alcohol use disorder show greater age-related decline of N-acetylaspartate in left dorsolateral prefrontal cortex. Drug Alcohol Depend. 2023 Jul 1;248:109901. doi: 10.1016/j.drugalcdep.2023.109901. Epub 2023 Apr 28. PMID 37146499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From 20MAR20-31AUG21 no participants were recruited due the mandatory hiatus of recruitment of human participants (forced by the COVID-19 pandemic) and the Principal Investigator's mobilization to active military service. The PI discussed the recruitment issues with the Stanford NeuroChoice Initiative funding agency, and it was decided to discontinue recruitment in JUL21.
Groups:
- Active iTBS; Sham iTBS: Intermittent theta burst transcranial magnetic stimulation: Participants will be randomized to active or sham iTBS conditions, and receive 20 iTBS sessions over the course of 2 weeks
Period: Overall Study
Arm/Group | Active iTBS | Sham iTBS
Started | 8 | 9
Completed | 5 | 7
Not Completed | 3 | 2
Not completed — Protocol Violation | 2 | 1
Not completed — Participant self-discharged against medical advice from treatment program during active study phase | 1 | 0
Not completed — Residential treatment team requested participant withdraw due to multiple conflicting appointments. | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active iTBS | Sham iTBS | Total
Number analyzed (Participants) | 8 | 9 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.0 (9.8) | 48.5 (12.4) | 42.3 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 8 | 8 | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 6 | 7 | 13
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 5 | 6 | 11
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 8 | 9 | 17
Education [Mean (Standard Deviation); unit: years] | 13.5 (1.5) | 13.3 (1.8) | 13.4 (1.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Were Abstinent Through Month 6
Description: Number of particiants in active vs. sham who maintained completed abstinence from alcohol/substance over 6 months post final rTMS session.
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Active iTBS | Sham iTBS
Number analyzed (Participants) | 8 | 9
Participants | 5 | 7
Statistical Analysis 1: Comparison: Active iTBS vs Sham iTBS; Test type: Other — Chi-Square comparison of frequencies; p = 0.99, Chi-squared — A p-value of <0.05 is considered statistically significant; Pearson Chi-Square = 0.17

2. Secondary Outcome: Left Dorsolateral Prefrontal Region Glutamate/Creatine Ratio
Description: Left dorsolateral prefrontal region glutamate/creatine ratio pre and post active/sham iTBS. Data were recorded in international units (IU) and converted to Z scores based on the entire sample (unit normal distribution, mean of 0, standard deviation of 1). Higher Z scores (standard deviation above the mean) indicate a greater metabolite concentration ratio and better functioning.
Time Frame: baseline and follow-up (approximately 2 weeks)
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Active iTBS | Sham iTBS
Number analyzed (Participants) | 4 | 7
z-score
  baseline | 0.31 (0.29) | 0.02 (0.30)
  week 2 | 0.25 (0.29) | 0.29 (0.22)
Statistical Analysis 1: Comparison: Active iTBS vs Sham iTBS; Linear mixed modeling; Test type: Other; p = 0.68, Mixed Models Analysis — p < .05 considered statistically significant; Slope = -0.20 — Rate of change compared between groups using linear mixed modeling

3. Secondary Outcome: Left Dorsolateral Prefrontal Cortex Thickness
Description: Left dorsolateral prefrontal cortex thickness pre and post active/sham iTBS; hypothesized that increased thickness corresponds to improved cytoarchitectural integrity of the left dorsolateral prefrontal cortex.
Time Frame: baseline and follow-up (approximately 2 weeks)
Population: Participants with data available at each respective assessment point.
Measure: Mean (Standard Deviation); unit: mm
Arm/Group | Active iTBS | Sham iTBS
Number analyzed (Participants) | 8 | 9
mm
  Baseline | 2.34 (0.14) | 2.36 (0.15)
  Follow-up: number analyzed (Participants) | 4 | 5
  Follow-up | 2.39 (0.17) | 2.37 (0.19)
Statistical Analysis 1: Comparison: Active iTBS vs Sham iTBS; Test type: Other; p = 0.34, Mixed Models Analysis — p-value < .05 considered statistically significant

4. Secondary Outcome: General Depressive Symptoms
Description: Beck Depression Inventory-II score pre and post active/sham iTBS (score range, 0 to 63, higher scores indicate more severe symptoms).
Time Frame: baseline and follow-up (approximately 2 weeks)
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active iTBS | Sham iTBS
Number analyzed (Participants) | 4 | 7
score on a scale
  Baseline | 18.4 (3.4) | 18.0 (3.1)
  Follow-up | 10.0 (4.0) | 11.9 (2.9)
Statistical Analysis 1: Comparison: Active iTBS vs Sham iTBS; Test type: Other — Linear mixed modeling; p = 0.70, Mixed Models Analysis — p < .05 considered statistically significant; Slope = -1.99 — Rate of change compared between groups using linear mixed modeling

5. Secondary Outcome: Anhedonic Depressive Symptoms
Description: Anhedonic depressive symptoms from Mood and Anxiety Symptom Questionnaire (MASQ, 30-item version; score range: 10 to 50, high scores correspond to more severe symptoms).
Time Frame: baseline and follow-up (approximately 2 weeks)
Population: Participants with available data are included in the analysis.
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Active iTBS | Sham iTBS
Number analyzed (Participants) | 4 | 8
score on a scale
  baseline | 29.1 (2.8) | 32.7 (2.6)
  Follow-up | 22.5 (3.3) | 30.5 (2.4)
Statistical Analysis 1: Comparison: Active iTBS vs Sham iTBS; Linear mixed modeling; Test type: Other; p = 0.11, Mixed Models Analysis — p < .05 considered statistically significant; Slope = 0.30

ADVERSE EVENTS:
Time Frame: Baseline through 6 months after conclusion of treatment
Description: Participants were systematically screened for any biomedical, psychiatric or other physical condition that was associated with serious adverse events or adverse events.
Arm/Group | Active iTBS | Sham iTBS
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/9
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9
Other Adverse Events (participants affected / at risk) | 0/8 | 0/9

LIMITATIONS AND CAVEATS:
The study was terminated early before enrolling the planned number of participants, therefore the data analysis is underpowered.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-08-01): https://cdn.clinicaltrials.gov/large-docs/31/NCT03291431/Prot_SAP_000.pdf
  • Informed Consent Form (2021-11-29): https://cdn.clinicaltrials.gov/large-docs/31/NCT03291431/ICF_001.pdf